CLINICAL TRIAL: NCT00002803
Title: COOPERATIVE MULTICENTER TRIAL FOR THE TREATMENT OF INFANTS WITH NEUROBLASTOMA
Brief Title: Combination Chemotherapy or Observation Following Surgery in Treating Infants With Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064903; GER-NB95-S; EU-96003
Record Dates: First submitted 1999-11-01; First posted 2004-05-12 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2008-04

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Cyclophosphamide; Doxorubicin; Vincristine

INTERVENTIONS:
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: vincristine sulfate
Procedure: conventional surgery

SUMMARY:
RATIONALE: Sometimes neuroblastoma will regress without treatment, but sometimes additional treatment may be necessary. Giving more than one chemotherapy drug after surgery to remove the tumor may kill more tumor cells.

PURPOSE: Phase II trial to study combination chemotherapy or observation following surgery in treating infants with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the incidence of spontaneous regression of localized neuroblastoma in infants. II. Determine how many infants with neuroblastoma do not need chemotherapy. III. Evaluate the time course of regression by radiologic criteria and catecholamine metabolites. IV. Determine the reliability of risk estimation by molecular characteristics (N-myc amplification, CD44, del 1p) compared to clinical criteria. V. Evaluate whether reduced therapeutic toxicity results in a decrease in treatment-related deaths. VI. Correlate cytostatic drug levels with chemotherapy side effects.

OUTLINE: All patients undergo resection of the primary tumor and N-myc determination within 6 months of age, unless critically ill, then are treated according to risk. Patients with amplified N-myc or with indeterminate N-myc amplification but with other risk features are treated per protocol GER-NB90. Stage 4S patients who are critically ill or thrombocytopenic receive doxorubicin, vincristine, and cyclophosphamide over 7 days. Patients with no amplification of N-myc are observed for 6 months (until between 12 and 18 months of age). Patients with minimal residual disease (less than 10% or diameter no greater than 2-5 mm) continue observation, while those with residual disease but no disease progression undergo repeat biopsy. Patients whose biopsy indicates tumor regression also continue observation. All other patients, including those with disease progression, are treated per protocol GER-NB90.

PROJECTED ACCRUAL: 36-44 patients per year will be accrued (22-27 patients with stages 1-3, 8-10 patients with stage 4S, and 6-7 patients with stage 4 neuroblastoma).

ELIGIBILITY:
DISEASE CHARACTERISTICS: See General Eligibility Criteria

PATIENT CHARACTERISTICS: See General Eligibility Criteria

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 1995-07; Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Berthold, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- University of Cologne, Frechen, Germany

REFERENCES:
- [Background] Hero B, Simon T, Spitz R, Ernestus K, Gnekow AK, Scheel-Walter HG, Schwabe D, Schilling FH, Benz-Bohm G, Berthold F. Localized infant neuroblastomas often show spontaneous regression: results of the prospective trials NB95-S and NB97. J Clin Oncol. 2008 Mar 20;26(9):1504-10. doi: 10.1200/JCO.2007.12.3349. PMID 18349403
- [Background] von Schweinitz D, Hero B, Berthold F. The impact of surgical radicality on outcome in childhood neuroblastoma. Eur J Pediatr Surg. 2002 Dec;12(6):402-9. doi: 10.1055/s-2002-36952. PMID 12548494
- [Result] Krams M, Hero B, Berthold F, Parwaresch R, Harms D, Rudolph P. Proliferation marker KI-S5 discriminates between favorable and adverse prognosis in advanced stages of neuroblastoma with and without MYCN amplification. Cancer. 2002 Feb 1;94(3):854-61. PMID 11857322